CLINICAL TRIAL: NCT01480089
Title: Surgical Pain Control With Ropivacaine by Atomized Delivery
Acronym: SPRAY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Elizabeth Mueller, Associate Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 203353
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Surgical Pain Management; Robotic surgery; Ropivacaine
MeSH Terms: conditions — Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomized Intraperitoneal Saline (AIS) (Placebo Comparator): Participants randomized to this arm will be given atomized intraperitoneal saline(AIS).
  Interventions: Drug: Atomized Intraperitoneal Saline (AIS)
- Intraperitoneal Ropivacaine(AIR) (Active Comparator): Participants randomized to this arm will receive atomized intraperitoneal ropivacaine (AIR).
  Interventions: Drug: Intraperitoneal Ropivacaine (AIR)

INTERVENTIONS:
Drug: Intraperitoneal Ropivacaine (AIR) — Ropivacaine 2 mg/kg per lean body mass up to no more than 200mg total dose will be atomized and delivered into the peritoneal cavity at the completion of surgery.
  Other Names: Ropivacaine
  Arms: Intraperitoneal Ropivacaine(AIR)
Drug: Atomized Intraperitoneal Saline (AIS) — Atomized saline will be administered to the peritoneal cavity at the completion of surgery.
  Other Names: Placebo
  Arms: Atomized Intraperitoneal Saline (AIS)

SUMMARY:
The purpose of this trial is to determine the effect of spraying a local anesthetic called Ropivacaine (numbing medicine) into the abdominal cavity prior to surgery. Ropivacaine is a local anesthetic used to block pain in the body. There are studies showing that Ropivacaine decreases the pain of surgery with minimally invasive (laparoscopic) appendix and gallbladder removal but has not been tried in robotic pelvic surgery.

DETAILED DESCRIPTION:
Practice guidelines from the American Society of Anesthesiologists peri-operative techniques for pain management have remained essentially unchanged over the last 10 years (3). Current acute pain-management strategies include 1.) Epidural or intrathecal opioids 2.) Patient-controlled devices delivering systemic opioids and 3.) Regional techniques such as peripheral nerve blocks and post-incisional infiltration with local anesthetics.

The use of epidural and systemic opioids results in significant side-effects such as post-operative nausea and ileus which often lead to increased hospital stay. The literature supporting the benefit of preincisional infiltration with anesthetics remains equivocal.

A recently published study describes the use of intraperitoneal Ropivacaine (2mh/kg) during laparoscopic appendectomy(4). The study was a randomized, double-blinded, placebo-controlled study using Ropivacaine (vs placebo) injected through the laparoscopic ports prior to the start of the appendectomy in 63 patients(4).

Patients treated with Ropivacaine had a significant decrease in visual analog pain scores post-operatively and had decreased narcotic use during their hospital stay compared to placebo. There were no side-effects found with the one-time use of the Ropivacaine.

The results of the above study and review of an additional 24 randomized controlled trials conducted from 1993-2003 are not felt to be generalizable to pelvic surgery where port placement and the operative procedures vary significantly. Hence this study was undertaken to investigate the role of intraperitoneal Ropivacaine as an adjuvant to muscle relaxants and narcotics at the time of pelvic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Consent to undergo robotic assisted gynecologic or urologic surgery
* Between the ages of 18 and 75
* Able to consent, fill out study documents, and complete all study procedures and follow-up visits

Exclusion Criteria:

* Patients with an allergy to local anesthetics
* Patients with severe underlying cardiovascular, renal or hepatic disease
* Pregnant patients

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Mueller, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available

REFERENCES:
- [Background] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Background] Hartog CS, Rothaug J, Goettermann A, Zimmer A, Meissner W. Room for improvement: nurses' and physicians' views of a post-operative pain management program. Acta Anaesthesiol Scand. 2010 Mar;54(3):277-83. doi: 10.1111/j.1399-6576.2009.02161.x. Epub 2009 Nov 12. PMID 19912126
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Boddy AP, Mehta S, Rhodes M. The effect of intraperitoneal local anesthesia in laparoscopic cholecystectomy: a systematic review and meta-analysis. Anesth Analg. 2006 Sep;103(3):682-8. doi: 10.1213/01.ane.0000226268.06279.5a. PMID 16931681
- [Background] Kang H, Kim BG. Intraperitoneal ropivacaine for effective pain relief after laparoscopic appendectomy: a prospective, randomized, double-blind, placebo-controlled study. J Int Med Res. 2010 May-Jun;38(3):821-32. doi: 10.1177/147323001003800309. PMID 20819419
- [Background] McClure JH. Ropivacaine. Br J Anaesth. 1996 Feb;76(2):300-7. doi: 10.1093/bja/76.2.300. No abstract available. PMID 8777115
- [Background] Bleckner LL, Bina S, Kwon KH, McKnight G, Dragovich A, Buckenmaier CC 3rd. Serum ropivacaine concentrations and systemic local anesthetic toxicity in trauma patients receiving long-term continuous peripheral nerve block catheters. Anesth Analg. 2010 Feb 1;110(2):630-4. doi: 10.1213/ANE.0b013e3181c76a33. Epub 2009 Dec 2. PMID 19955504
- [Background] Labaille T, Mazoit JX, Paqueron X, Franco D, Benhamou D. The clinical efficacy and pharmacokinetics of intraperitoneal ropivacaine for laparoscopic cholecystectomy. Anesth Analg. 2002 Jan;94(1):100-5, table of contents. doi: 10.1097/00000539-200201000-00019. PMID 11772809
- [Background] Mueller ER, Kenton K, Anger JT, Bresee C, Tarnay C. Cosmetic Appearance of Port-site Scars 1 Year After Laparoscopic Versus Robotic Sacrocolpopexy: A Supplementary Study of the ACCESS Clinical Trial. J Minim Invasive Gynecol. 2016 Sep-Oct;23(6):917-21. doi: 10.1016/j.jmig.2016.05.001. Epub 2016 May 12. PMID 27180224
- [Derived] Collins GG, Gadzinski JA, Fitzgerald GD, Sheran J, Wagner S, Edelstein S, Mueller ER. Surgical Pain Control With Ropivacaine by Atomized Delivery (Spray): A Randomized Controlled Trial. J Minim Invasive Gynecol. 2016 Jan;23(1):40-5. doi: 10.1016/j.jmig.2015.07.018. Epub 2015 Aug 1. PMID 26241686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women undergoing minimally invasive laparoscopic surgery in urogynecology, benign gynecology, and gynecologic-oncology clinics were recruited. All women who were scheduled to undergo a minimally invasive hysterectomy for benign and cancerous conditions between February 2012 and March 2013 were invited to participate.
Pre-assignment Details: One enrolled participant was excluded from the trial before assignment to groups because her physician prescribed Ropivacaine and, consequently, the participant was converted to open label before study drug was assigned or administered.
Groups:
- Atomized Intraperitoneal Saline (AIS): Participants randomized to this arm are given atomized intraperitoneal saline(AIS) to the peritoneal cavity at the completion of surgery.
- Intraperitoneal Ropivacaine(AIR): Participants randomized to this arm receive atomized intraperitoneal ropivacaine (AIR). That is, 2 mg/kg of lean body mass up to no more than 200mg total dose is atomized and delivered into the peritoneal cavity at the completion of surgery.
Period: Overall Study
Arm/Group | Atomized Intraperitoneal Saline (AIS) | Intraperitoneal Ropivacaine(AIR)
Started | 25 | 30
Completed | 25 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All women randomized to treatment were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intraperitoneal Ropivacaine(AIR) | Atomized Intraperitoneal Saline (AIS) | Total
Number analyzed (Participants) | 25 | 30 | 55
Age, Continuous [Mean (Full Range); unit: years] | 54.6 [31 to 72] | 58.8 [31 to 74] | 56.9 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 21 | 22 | 43
  Black | 2 | 5 | 7
  Hispanic | 1 | 2 | 3
  Asian | 1 | 1 | 2
Surgical Approach [Number; unit: participants]
  Laparoscopic | 11 | 11 | 22
  Robotic | 14 | 19 | 33
Attending Specialty [Number; unit: participants]
  Benign Gynecology | 2 | 4 | 6
  Urogynecology | 12 | 14 | 26
  Gynecologic Oncology | 11 | 12 | 23
Length of Hospital Stay [Number; unit: participants]
  Less than 24 hours | 0 | 0 | 0
  24 to 48 hours | 19 | 23 | 42
  Greater than 48 hours | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Post-op Pain With Atomized Intraperitoneal Ropivacaine (AIR)
Description: Participants are asked to rate their pain level using the visual analog scale (VAS). The VAS is a measurement of pain where respondents specify their level of pain by indicating a position along a continuous line between two end-points. The VAS used in this study was a horizontal line of 100 mm length anchored by two word descriptors - one word at each end: No pain (left end) and Very Severe Pain (right end). The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks. The VAS range is 0 to 100.
Time Frame: 2 hours after surgery
Population: All individuals randomized are included in this analysis.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intraperitoneal Ropivacaine(AIR) | Atomized Intraperitoneal Saline (AIS)
Number analyzed (Participants) | 25 | 30
millimeters | 2.536 (2.7) | 3.844 (3.0)
Statistical Analysis 1: Comparison: Intraperitoneal Ropivacaine(AIR) vs Atomized Intraperitoneal Saline (AIS); The null hypothesis is that the mean VAS score 2 hours post surgery is equivalent for individuals randomized to Intraperitoneal Ropivacaine(AIR) and those randomized to Atomized Intraperitoneal Saline (AIS); Test type: Superiority or Other; p = .098, t-test, 2 sided; Mean Difference (Final Values) = -1.308, 95% CI 2-sided [-2.830 to 0.214], Standard Error of Mean 0.777

2. Secondary Outcome: Post-op Pain With Atomized Intraperitoneal Ropivacaine (AIR)
Description: as for outcome 1
Time Frame: 12 hours after surgery
Population: All individuals randomized are included in this analysis.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Intraperitoneal Ropivacaine(AIR) | Atomized Intraperitoneal Saline (AIS)
Number analyzed (Participants) | 25 | 30
millimeters | 2.154 (1.9) | 2.219 (2.00)
Statistical Analysis 1: Comparison: Intraperitoneal Ropivacaine(AIR) vs Atomized Intraperitoneal Saline (AIS); The null hypothesis is that the mean VAS score 12 hours post surgery is equivalent for individuals randomized to Intraperitoneal Ropivacaine(AIR) and those randomized to Atomized Intraperitoneal Saline (AIS); Test type: Superiority or Other; p = .90, t-test, 2 sided; Mean Difference (Final Values) = -0.065, 95% CI 2-sided [-1.103 to 0.973], Standard Error of Mean 0.530

ADVERSE EVENTS:
Time Frame: Adverse event data were collected between August 19, 2011 and February 20, 2013 (1 year, 6.1 months)
Arm/Group | Intraperitoneal Ropivacaine(AIR) | Atomized Intraperitoneal Saline (AIS)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/30
Other Adverse Events (participants affected / at risk) | 0/25 | 0/30

LIMITATIONS AND CAVEATS:
There are no caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes